CLINICAL TRIAL: NCT05704946
Title: The Effect of Lavender Inhalation on Sleep Quality in Individuals With Coronary Heart Disease: a Randomized Controlled Study
Brief Title: The Effect of Lavender Inhalation on Sleep Quality in Individuals With Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sevgi Deniz Dogan, assistant professor, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 5312256930
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Nursing Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): The patients will be given a standard brand of lavender oil by the researcher, and they will be informed about how to use it (they should drop 2 drops of lavender oil on the right side of their pillow and 2 drops on the left side of their pillow every evening for a month after discharge).
  Interventions: Other: THE EFFECT OF LAVENDER INHALATION ON SLEEP QUALITY IN INDIVIDUALS WITH CORONARY HEART DISEASE
- control group (No Intervention): Standard care will be applied.

INTERVENTIONS:
Other: THE EFFECT OF LAVENDER INHALATION ON SLEEP QUALITY IN INDIVIDUALS WITH CORONARY HEART DISEASE — The index includes 24 questions that evaluate the quality of sleep and the type and severity of sleep disorders experienced in the last 1 month period. The total score in the index takes a value between 0-21. If the total score is higher than 5, it is interpreted as poor sleep quality.
  Arms: experiment group

SUMMARY:
The study is planned to be conducted as a two-group randomized controlled trial to determine the effect of lavender inhalation on individuals with coronary heart disease. Research data will be collected at Çukurova University Medical Faculty Balcalı Hospital Cardiology Clinic between January-June 2023. In the study, at least 56 samples were found to be sufficient for the sample size. The data of the study will be collected using the Personal Information Form and the Pittsburg Sleep Quality Index.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and speak Turkish,
* Who agreed to participate in the research

Exclusion Criteria:

* People with communication difficulties and mental retardation
* People with coagulation disorders
* People with migraines and chronic headaches
* People with an allergy to lavender (Lavandula angustifolia Mill)
* It is the desire to leave the research.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Effect of lavender inhalation on sleep quality | one months
  The index includes 24 questions that evaluate the quality of sleep and the type and severity of sleep disorders experienced in the last 1 month period. The total score in the index takes a value between 0-21. If the total score is higher than 5, it is interpreted as poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Çukurova University Institute of Health Sciences, Adana, Turkey (Türkiye)